CLINICAL TRIAL: NCT04803383
Title: The Effects of Tele-Yoga in Ankylosing Spondylitis Patients: A Randomized Controlled Trial
Brief Title: The Effects of Tele-Yoga in Ankylosing Spondylitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Yasemin ACAR, Research assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/05-34
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Ankylosing Spondylitis; Yoga
Keywords: ankylosing spondylitis; yoga
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Yoga Group (Experimental): Patients in the tele-yoga group will participate in tele-yoga sessions with a maximum of 5 people in each group by video-conference method for 8 weeks, 3 days a week. Assessments will perform just before starting to study and after the 8-week tele-yoga program
  Interventions: Other: Tele-yoga
- Control group (No Intervention): Patients in the waiting list control group will be asked to continue their normal physical activities during the 8-week study, not to start a new exercise program, and to report any changes in the drug or dosage used. Control group's assessments will be performed when they are included in the study and at the end of 8 weeks. After these assessments, patients who wish will participate in the tele-yoga program.

INTERVENTIONS:
Other: Tele-yoga — Tele-yoga training 3 days a week for 8 weeks
  Arms: Tele-Yoga Group

SUMMARY:
The aim of this study is to investigate the effect of tele-yoga on functional level, disease activity, spinal mobility, balance, aerobic capacity, sleep quality, anxiety, depression, stress, mindfulness and quality of life in patients with ankylosing spondylitis

DETAILED DESCRIPTION:
Yoga is an ancient discipline that emerged in India thousands of years ago, designed to bring balance and health to the physical, mental, emotional and spiritual dimensions of the individual.Due to its therapeutic effects, yoga can be considered as an alternative approach for those with rheumatic disease. Because of Covid-19, which has changed the world and the lifestyle of people, tele-yoga practice can be considered as an alternative instead of traditional face-to-face yoga classes. The use of online platforms provides a good environment for yoga training at home. The aim of this study is to investigate the effects of tele-yoga on functional level, disease activity, spinal mobility, balance, sleep quality, depression, mindfulness and quality of life in patients with ankylosing spondylitis.

60 AS patients who meet the inclusion criteria will be assigned to the tele-yoga or waiting list control group by the block randomization method. Patients in the tele-yoga group will participate in tele-yoga sessions with a maximum of 5 people in each group by video-conference method for 8 weeks, 3 days a week. Assessments will perform just before starting to study and after the 8-week tele-yoga program. Patients in the waiting list control group will be asked to continue their normal physical activities during the 8-week study, not to start a new exercise program, and to report any changes in the drug or dosage used. Control group's assessments will be performed when they are included in the study and at the end of 8 weeks. After these assessments, patients who wish will participate in the tele-yoga program.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis(AS) patients diagnosed according to modified New York criteria
* To be volunteer
* To have the necessary equipment to provide internet access and connection

Exclusion Criteria:

* Presence of systemic, orthopedic neurological or cognitive disease other than ankylosing spondylitis
* Regular exercise in the last 3 months
* Pregnancy
* Not attending 4 consecutive yoga sessions
* Changing the drug during the study
* Has an acute attack during the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Functional Index (BASFI) | Change from Baseline at 8 weeks
  Assess functional capacity. This self-assessment instrument consists of eight specific questions regarding function in AS and two questions reflecting the patient's ability to cope with everyday life regarding function in AS and two questions reflecting the patient's ability to cope with everyday life.The BASFI score is calculated by dividing the sum of the scores from 10 questions by 10. Score range is 0-10, with 0 reflecting no functional impairments and 10 reflecting maximal impairment.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Spinal Metrology Index (BASMI) | Change from Baseline at 8 weeks
  Asses spinal mobility. The total score ranges from 0 to 10. Higher scores mean poor spinal mobility.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Change from Baseline at 8 weeks
  Assess disease activity. The total score ranges from 0 to 10. High scores mean an increase in disease activity.
Assessment of Spondyloarthritis international Society Health Index (ASAS HI) | Change from Baseline at 8 weeks
  The ASAS HI contains 17 items (dichotomous response option: 'I agree' and 'I do not agree') addressing different aspects of functioning. The total ASAS HI score is between 0 and 17. Lower score indicates a better and a higher score indicates an inferior health status
Muscular endurance: | Change from Baseline at 8 weeks
  Sit-up and push-up tests will be used to evaluate muscular endurance.
Balance | Change from Baseline at 8 weeks
  Balance performance will be assessed by the Balance Master System (NeuroCom® International Inc., USA).
Aerobic Capacity | Change from Baseline at 8 weeks
  The incremental Shuttle Walk Test will be used to determine aerobic capacity
Pittsburgh Sleep Quality Index | Change from Baseline at 8 weeks
  Assess quality of sleep
The Hospital Anxiety And Depression Scale(HADS) | Change from Baseline at 8 weeks
  The HADS is a 14-item self-report questionnaire that measures anxiety (7 items) and depression (7 items) symptoms.
Stress | Change from Baseline at 8 weeks
  Stress will be assessed with Perceived Stress Scale (PSS).The scale consists of 14 items and total score ranges from 0 to 56. High scores indicate high stress perception.
Mindfulness | Change from Baseline at 8 weeks
  Mindful Attention Awareness Scale will be used. The scale consists of 15 items. The total score that can be obtained from the scale is between 15 and 90. High scores reflect more mindfulness.
Short Form-36 (SF-36) | Change from Baseline at 8 weeks
  Assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: YASEMİN ACAR, Principal Investigator — Dokuz Eylul University; NURSEN İLÇİN, Study Director — Dokuz Eylul University; İSMAİL SARI, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acar Y, Ilcin N, Sari I. The Effects of Tele-Yoga in Ankylosing Spondylitis Patients: A Randomized Controlled Trial. J Integr Complement Med. 2023 Nov;29(11):727-737. doi: 10.1089/jicm.2023.0022. Epub 2023 May 31. PMID 37257184